CLINICAL TRIAL: NCT06434714
Title: Management of Postoperative Pain After Cesarean Delivery Using Bridge Auricular Percutaneous Nerve Field Stimulator
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Inova Health Care Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INOVA-2023-131
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Post-operative Pain, Acute; Cesarean Section; Opioid Use Disorder; Opioids; Harmful Use
Keywords: cesarean section; post-operative pain; opioid abuse; non-pharmacologic therapy
MeSH Terms: conditions — Pain, Postoperative; Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: Double-blinded, placebo-controlled, 3 arm randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will be randomized to either active Bridge device, sham (non-functional) device, or standard of care post-operative pain regimen. Participants, care providers, and investigators will be blinded to those in active or sham device groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Bridge device (Active Comparator): Bridge device placed in post-anesthesia care unit (PACU) and worn until end-of-life of the device (at 5 days) in addition to standard of care pain medications as per institutional policy
  Interventions: Device: Auricular percutaneous nerve field stimulator
- Sham device (Sham Comparator): Sham (non-functional) Bridge device placed in post-anesthesia care unit (PACU) and worn until 5 days post-delivery in addition to standard of care pain medications as per institutional policy
  Interventions: Device: Sham auricular percutaneous nerve field stimulator
- Standard of care (No Intervention): Standard of care pain medications only as per institutional policy

INTERVENTIONS:
Device: Auricular percutaneous nerve field stimulator — Percutaneous nerve field stimulator device placed on the ear for 5 days
  Other Names: Bridge
  Arms: Bridge device
Device: Sham auricular percutaneous nerve field stimulator — Non-functioning percutaneous nerve field stimulator device placed on the ear for 5 days
  Arms: Sham device

SUMMARY:
Post-cesarean section (CS) pain is commonly treated with acetaminophen, ibuprofen, and opioid medications as needed following delivery. About 300,000 women annually who were exposed to opioids after CS will go on to use opioids chronically. Reducing the quantity of post-CS opioids has been shown to decrease the amount of opioids used without compromising pain control. Bridge is a small device that sits on the outer ear and works similarly to a transcutaneous electrical nerve stimulation (TENS) unit to decrease pain sensation without medications. It has been shown to effectively reduce pain to decrease medication requirements after surgeries. This study aims to see if women receiving the Bridge device use need less pain medication than those without the device.

DETAILED DESCRIPTION:
Cesarean delivery is one of the most performed surgeries in the U.S. with approximately 1.15 million surgeries performed annually. Despite this, postoperative pain management remains a challenge. Prescribed total milligram morphine equivalents (MMEs) can range from 25 MMEs (equivalent to 3.3 oxycodone 5-mg tablets) to 1,950 MMEs (equivalent to 260 oxycodone 5-mg tablets). Additionally, the post discharge analgesia prescription is not correlated with the 24-hour predischarge opioid use or pain score. Most U.S. women who are prescribed opioids after a cesarean delivery receive at least 10 more tablets than necessary. A study looking at individualizing opioid prescriptions based on inpatient requirements found that women used about 60% of their prescription, regardless of the amount of opioids prescribed. Decreasing opioid requirement after cesarean delivery, can decrease women's exposure to opioids, reduce the risk of neonatal central nervous system depression due to exposure in breastmilk, and limit the potential for extra opioids from unused, filled prescriptions to fall into the wrong hands. Post-cesarean mothers use opioids for a median of 8 days after delivery. Bridge is a minimally invasive device shown in previous studies to reduce pain medication requirements in the post-operative acute recovery period. The device is a auricular percutaneous electrical nerve stimulator that modulates pain receptors leading to reduced pain sensation. This trial study to examine the utility of the Bridge device as an adjunct to standard of care post-cesarean pain regimens (acetaminophen, ibuprofen or ketorolac, and oxycodone or other similar opioid). Post-cesarean patients will be randomized in a 1:1:1 ratio to Bridge device, sham device, or standard of care treatment and followed through the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Female 18 years or older able to provide informed consent in English or Spanish.
* Scheduled for cesarean delivery under neuraxial anesthesia.
* Intact skin surface behind and around the ear at the site of electrode application.

Exclusion Criteria:

* Active drug abuse.
* Chronic opioid user.
* Severe chronic pain.
* Hemophilia.
* Cardiac pacemaker or implantable electronic devices.
* Psoriasis vulgaris or other skin conditions precluding safe device application.
* Previous history of sensitivity to compound benzoin tincture.
* Hearing aid precluding proper placement of the device or removing which interferes with their hearing ability.
* Subject is concurrently participating in another research study with an investigational drug or medical device that in the Investigator's opinion could impact subject safety or study results.
* Subject with reasons to maintain an epidural beyond operative room.
* Subject with complex surgery or subject who may need more than a cesarean surgery with possible tubal sterilization procedure.
* Subject is deemed not suitable for the study at the discretion of the principal Investigator.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Total opioid intake on post-operative day 4 | Four days
  Total opioid intake in morphine milligram equivalents (MME) on post-operative day 4

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Saad, MD, Principal Investigator — Inova Health Systems; Ellen M Murrin, DO, Principal Investigator — Inova Health Systems
Locations (1):
- Inova Fairfax Medical Campus, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osmundson SS, Min JY, Grijalva CG. Opioid prescribing after childbirth: overprescribing and chronic use. Curr Opin Obstet Gynecol. 2019 Apr;31(2):83-89. doi: 10.1097/GCO.0000000000000527. PMID 30789842
- [Background] Bateman BT, Franklin JM, Bykov K, Avorn J, Shrank WH, Brennan TA, Landon JE, Rathmell JP, Huybrechts KF, Fischer MA, Choudhry NK. Persistent opioid use following cesarean delivery: patterns and predictors among opioid-naive women. Am J Obstet Gynecol. 2016 Sep;215(3):353.e1-353.e18. doi: 10.1016/j.ajog.2016.03.016. Epub 2016 Mar 17. PMID 26996986
- [Background] Chelly JE, Monroe AL, Planinsic RM, Tevar A, Norton BE. Auricular field nerve stimulation using the NSS-2 BRIDGE(R) device as an alternative to opioids following kidney donor surgery. J Complement Integr Med. 2021 Nov 1;19(2):449-454. doi: 10.1515/jcim-2021-0208. eCollection 2022 Jun 1. PMID 34714990
- [Background] Lim G, LaSorda KR, Monroe AL, Chelly JE. Auricular percutaneous nerve field stimulator device as alternative therapy for Cesarean delivery analgesia: proof of concept. Can J Anaesth. 2019 Dec;66(12):1522-1523. doi: 10.1007/s12630-019-01465-x. Epub 2019 Aug 20. No abstract available. PMID 31432323